CLINICAL TRIAL: NCT02600741
Title: A 12-Month Randomized, Open-Label Study of Caregiver Psycho-education and Skills Training in Patients Recently Diagnosed With Schizophrenia, Schizoaffective Disorder, or Schizophreniform Disorder and Receiving Paliperidone Palmitate or Oral Antipsychotic Treatment
Brief Title: Family Intervention in Recent Onset Schizophrenia Treatment (FIRST)
Acronym: FIRST
Status: Completed | Type: Observational
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR106399; R092670SCH4043 (Other: Janssen Scientific Affairs)
Record Dates: First submitted 2015-09-29; First posted 2015-11-09 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Caregiver; Psycho-education and skills training; Paliperidone Palmitate; Oral Antipsychotic
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Chlorpromazine; Droperidol; Fluphenazine; Haloperidol; Loxapine; Perphenazine; Pimozide; Prochlorperazine; Thiothixene; Thioridazine; Trifluoperazine; Aripiprazole; asenapine; Clozapine; iloperidone; Olanzapine; Quetiapine Fumarate; Risperidone; ziprasidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group 1: Caregivers randomized to this group will receive up to 16 sessions of study-provided caregiver psycho-education and skills training sessions they are able to attend within a 6-month period. Each patient will be paired with a caregiver and patients will continue their routine antipsychotic treatments prescribed by their treating physician.
  Interventions: Other: Caregiver psycho-education and skills training; Drug: Paliperidone palmitate; Drug: Chlorpromazine; Drug: Droperidol; Drug: Fluphenazine; Drug: Haloperidol; Drug: Loxapine; Drug: Perphenazine; Drug: Pimozide; Drug: Prochlorperazine; Drug: Thiothixene; Drug: Thioridazine; Drug: Trifluoperazine; Drug: Aripiprazole; Drug: Asenapine; Drug: Clozapine; Drug: Iloperidone; Drug: Olanzapine; Drug: Paliperidone; Drug: Quetiapine; Drug: Risperidone; Drug: Ziprasidone
- Study group 2: Caregivers randomized to this group will receive whatever caregiver support that is customarily available at the study site, if any. Each patient will be paired with a caregiver and patients will continue their routine antipsychotic treatments prescribed by their treating physician.
  Interventions: Other: Caregiver support available at the study site; Drug: Paliperidone palmitate; Drug: Chlorpromazine; Drug: Droperidol; Drug: Fluphenazine; Drug: Haloperidol; Drug: Loxapine; Drug: Perphenazine; Drug: Pimozide; Drug: Prochlorperazine; Drug: Thiothixene; Drug: Thioridazine; Drug: Trifluoperazine; Drug: Aripiprazole; Drug: Asenapine; Drug: Clozapine; Drug: Iloperidone; Drug: Olanzapine; Drug: Paliperidone; Drug: Quetiapine; Drug: Risperidone; Drug: Ziprasidone

INTERVENTIONS:
Other: Caregiver psycho-education and skills training — Caregivers will receive up to 16 sessions of study-provided caregiver psycho-education and skills training sessions they are able to attend within a 6-month period.
  Groups: Study group 1
Other: Caregiver support available at the study site — Caregivers will receive whatever caregiver support that is customarily available at the study site, if any.
  Groups: Study group 2
Drug: Paliperidone palmitate — Patients enrolled in this study will continue to receive routine treatment of paliperidone palmitate, as directed by their treating physician.
Drug: Chlorpromazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Droperidol — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Fluphenazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Haloperidol — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Loxapine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Perphenazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Pimozide — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Prochlorperazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Thiothixene — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Thioridazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Trifluoperazine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Aripiprazole — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Asenapine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Clozapine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Iloperidone — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Olanzapine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Paliperidone — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Quetiapine — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Risperidone — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.
Drug: Ziprasidone — Patients enrolled in this study will continue to receive routine treatment of oral antipsychotics, as directed by their treating physician.

SUMMARY:
The primary purpose of this study is to evaluate the overall effect of caregivers receiving a study-provided caregiver psycho-education and skills training program on the number of treatment failures (psychiatric hospitalization, psychiatric emergency room (ER) visit, crisis center visit, mobile crisis unit intervention, arrest/incarceration, and suicide or suicide attempt) in patients under their care during a 12 month period.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel group study of patients with schizophrenia, schizoaffective disorder, or schizophreniform disorder and their caregivers. Study will consist of a paired patient and caregiver. Patients will receive routine treatment, which may include oral antipsychotics or paliperidone palmitate, as directed by their treating physician. Caregivers for patients whose routine treatment is paliperidone palmitate will be randomized to receive either a study-provided caregiver psycho-education and skills training or usual caregiver support. Caregivers for patients whose routine treatment is oral antipsychotics will be randomized to the same Study Groups: Study Group 1: Study-provided caregiver psycho-education and skills training. Study Group 2: Usual caregiver support (caregiver support that is customarily provided by the study site, if any). Patients-caregiver pairs will be followed for up to 12 months following baseline assessment. Cumulative number of treatment failures over 12 months will be assessed primarily.

ELIGIBILITY:
Inclusion Criteria:

A) Caregivers

* Each caregiver must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate for the duration of the study
* Caregiver is able to have verbal interaction with the patient with schizophrenia, schizoaffective disorder, or schizophreniform disorder at least twice a week, per self-report

B) Patients

* Patients must have a clinical diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder made by a clinician with understanding of the Diagnostic and Statistical Manual of Mental Disorders (DSM V) criteria for these disorders
* Patients must be receiving ongoing psychiatric treatment at the study site and must be receiving oral antipsychotics or paliperidone palmitate long acting therapy

Exclusion Criteria:

* A) Caregivers
* Caregiver is mentally or physically incapable of adequately performing the required study procedures, as determined by the treatment team
* Caregiver has received structured or manualized psycho-education or skills training within 1 year prior to Screening B) Patients
* Patient is hospitalized (medical or psychiatric), incarcerated, or otherwise institutionalized at time of randomization
* Patient is considered to have significant potential for imminent harm to self and/or others as based on the judgment of the treatment team
* Patient is receiving assertive community treatment (ACT) or other high intensity case management services to prevent hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will consist of a paired patient and caregiver. A caregiver is defined as a person who has accepted responsibility for providing the patient with both assistance with activities of daily living and protection from harm. The patient will have a diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder.
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Number of Treatment Failures Over 12 Months | 12 months
  Treatment failure is defined as any of the following:
  1. Psychiatric hospitalization
  2. Psychiatric emergency room (ER) visit
  3. Crisis center visit
  4. Mobile crisis unit intervention
  5. Arrest/Incarceration
  6. Suicide or suicide attempt.

SECONDARY OUTCOMES:
Caregiver Burden Based on Involvement Evaluation Questionnaire (IEQ) Total Score at Month 12 | Month 12
  The IEQ is designed to measure levels of caregiver consequences among family members and friends of patients with schizophrenia. The 31 items included in this scale are answered on a 5 point Likert response scale and address consequences among 4 dimensions (tension, supervision, worrying, and urging).
Number of Treatment Failures in Patients Taking Oral Antipsychotics | 12 months
  Treatment failure is defined as any of the following:
  1. Psychiatric hospitalization
  2. Psychiatric emergency room (ER) visit
  3. Crisis center visit
  4. Mobile crisis unit intervention
  5. Arrest/Incarceration
  6. Suicide or suicide attempt.
Number of Treatment Failures in Patients Taking Paliperidone Palmitate | 12 months
  Treatment failure is defined as any of the following:
  1. Psychiatric hospitalization
  2. Psychiatric emergency room (ER) visit
  3. Crisis center visit
  4. Mobile crisis unit intervention
  5. Arrest/Incarceration
  6. Suicide or suicide attempt.
Patient Recovery Based on Total Illness Management and Recovery (IMR) Score | Month 6 and Month 12
  The IMR program was developed in order to help patients with schizophrenia or major mood disorders learn how to manage their illnesses more effectively in the context of pursuing their personal goals.
Change From Baseline in Clinical Global Impression - Severity (CGI-S) at Month 12 | Month 12
  The CGI-S rating scale is used to rate the severity of a patient's overall clinical condition on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) to 7 (amongst the most severely ill patients).
Change From Baseline in 12- Item Short Form Health Survey (SF-12) at Month 12 | Month 12
  The 12-item Short Form Health Survey (SF-12) is a self-administered, generic, 12-item questionnaire designed to cover the same 8 domains of functional health status and well-being included in the longer 36-item Short Form Health Survey (SF 36): physical functioning, role limitations due to physical health problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Chair — Janssen Scientific Affairs, LLC
Locations (34):
- United States (34):
  - Bullhead City, Arizona
  - Oceanside, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Lauderdale Lakes, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Orange City, Florida
  - Tallahassee, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Granite City, Illinois
  - Lombard, Illinois
  - Springfield, Illinois
  - Bloomington, Indiana
  - Lawrenceburg, Indiana
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Mount Pleasant, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - New York, New York
  - Staten Island, New York
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Eugene, Oregon
  - Lincoln, Rhode Island
  - Nashville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richland, Washington
  - Spokane, Washington

REFERENCES:
- [Derived] Mueser KT, Achtyes ED, Gogate J, Mancevski B, Kim E, Starr HL. Telehealth-Based Psychoeducation for Caregivers: The Family Intervention in Recent-Onset Schizophrenia Treatment Study. JMIR Ment Health. 2022 Apr 15;9(4):e32492. doi: 10.2196/32492. PMID 35436231